CLINICAL TRIAL: NCT06037772
Title: The Effect of Using Digital Games on Learning Satisfaction and Self-confidence in Providing Nursing Students With Subcutaneous Injection Skills
Brief Title: The Effect of Digital Game Use in Teaching Subcutaneous Injection Administration Skills to Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Burcu Demircan, Lecturer, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Bvu_Nursing-2
Record Dates: First submitted 2023-08-28; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Nursing Education
Keywords: learning satisfaction; self-confidence; digital game; nursing students
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: pretest-posttest, randomized controlled experimental design with experimental and control groups
Who Masked: Participant, Investigator
Masking Description: Informed consent form was obtained from the participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subcutaneous injection practice game (Experimental): After the subcutaneous injection was explained to the experimental group, the digital game developed for subcutaneous injection was explained and they were allowed to play the game for a week. Afterwards, the experimental group was shown the subcutaneous injection application on a low-reality model of the abdomen, and the students were allowed to practice the skill.
  Interventions: Other: subcutaneous injection administration game; Other: control group
- Traditional education (Active Comparator): The students in the control group were given the traditional education method (subcutaneous injection application on a low-reality abdominal model after the completion of the theoretical course on the subject of subcutaneous injection).
  Interventions: Other: control group

INTERVENTIONS:
Other: subcutaneous injection administration game — The subcutaneous injection practice game was developed to examine nursing students' injection practice skills and its effect on their satisfaction with learning.
  Arms: Subcutaneous injection practice game
Other: control group — only

SUMMARY:
The goal of this to determine the effect of a digital game-based application on learning satisfaction and self-confidence in the acquisition of subcutaneous drug administration skills by nursing students.

The research hypotheses it aims to answer are:

* Hypothesis 1: The subcutaneous injection knowledge level of the students who are educated with the digital game method is higher than the students who receive the traditional education.
* Hypothesis 2: The subcutaneous injection skill test scores of the students who were educated with the digital game method were higher than the students who received the traditional education.
* Hypothesis 3: The satisfaction and self-confidence level of the students who are educated with the digital game method towards subcutaneous injection is higher than the students who receive the traditional education.

DETAILED DESCRIPTION:
In studies on the use of digital games in nursing education; Students value instant feedback, visuals and experiential learning, the game developed to improve their decision-making and reasoning skills is extremely useful, useful and enjoyable, from nursing students to those with no previous operating room experience. It has been stated that when the application is made with a game-like simulation, the information is more permanent, they behave more collaboratively, and they experience less fear. The study was planned in a randomized controlled experimental design with pretest-posttest, experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Being a 1st year nursing student

Exclusion Criteria:

* Previous training in subcutaneous application skills

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Digital game method and subcutaneous injection knowledge level-pre-test | "1 week"
  The level of knowledge about subcutaneous injection was measured by the "Subcutaneous Injection Knowledge Test", which was prepared by the researchers in line with the literature and submitted to expert opinion and whose Content Validity was calculated. The subcutaneous injection knowledge test is a multiple choice test consisting of 25 questions. The scores obtained from the test will not be classified according to the level of achievement, the averages of the achievement scores of the groups were compared.
Digital game and subcutaneous injection skill level | "2 week"
  Subcutaneous injection skill level was measured with the "Subcutaneous Heparin Injection Administration Skill Checklist", which was prepared by the researchers in line with the literature and submitted to expert opinion and whose Content Validity was calculated. There are 33 items in the Subcutaneous Heparin Injection Administration Skill Checklist. Each item consists of three points as "adequate", "developmental" and "inadequate", respectively. The scores of these degrees are "2", "1", "0", respectively. The highest score that can be obtained from the test is "66" and the lowest score is "0".
Level of satisfaction and self-confidence in digital gaming and learning | "2 week"
  Students' satisfaction and self-confidence levels were measured with the Turkish validity and reliability study "Learning Satisfaction and Confidence in Learning Scale". The scale consists of "13" items and the 13th item of the scale is reverse coded. Each item was scored on a five-point Likert scale between "strongly disagree-strongly agree". The lowest score that can be obtained from the scale is 13, and the highest score is 65.

SECONDARY OUTCOMES:
Digital game method and subcutaneous injection knowledge level-post-test | "4 week"
  The level of knowledge about subcutaneous injection was measured by the "Subcutaneous Injection Knowledge Test", which was prepared by the researchers in accordance with the literature and presented to the expert opinion and whose Content Validity was calculated. The subcutaneous injection knowledge test is a multiple choice test consisting of 25 questions. The post-test was administered to both groups 2 weeks after all the interventions. The scores obtained from the test will not be classified according to the level of success, the averages of the groups' achievement scores will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Kaya, Professor, Study Director — İstanbul University-Cerrahpasa
Locations (1):
- Burcu Demircan, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Since the study phases have not yet been completed and the thesis process is ongoing, the data is not suitable for sharing.

DOCUMENTS (1):
  • Informed Consent Form (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT06037772/ICF_000.pdf